CLINICAL TRIAL: NCT03282422
Title: Effectiveness of the Functional Hand Splint and Specific Tasks in the Domiciliary Environment Applied to Children With Unilateral Cerebral Palsy. Randomized Clinical Trial
Brief Title: Effectiveness of the Functional Hand Splint and Specific Tasks in the Domiciliary Environment Applied to Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Collaborators: AIDIMO Asociación para la investigación en la discapacidad motriz (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF_TE_01_Versión 3
Record Dates: First submitted 2017-09-06; First posted 2017-09-14 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-04

CONDITIONS: Hemiplegia and Hemiparesis; Cerebral Palsy Infantile
Keywords: Cerebral palsy; Hemiplegia; Upper-limb splint; Home-based; Social Participation
MeSH Terms: conditions — Hemiplegia; Paresis; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Upper-limb splint and home-based protocol in specific tasks
  Interventions: Device: Home-based protocol in specific tasks; Device: Upper-limb splint
- Control group (Active Comparator): Home-based protocol in specific tasks
  Interventions: Device: Home-based protocol in specific tasks

INTERVENTIONS:
Device: Home-based protocol in specific tasks — The home-based protocol in specific tasks will be an individualized protocol designed for the child according to the results of the baseline assessment and will require active participation. It is a program that is integrated into the daily routines of the child. A study investigator will tell the family the procedure to follow.
Device: Upper-limb splint — In the case that treatment with splint is also received, a researcher of this study will take measurements of the hand and will provide the appropriate splint. The intensity of the application will be 5 days a week from monday to friday, for 6 hours a day, for a period of 6 weeks.
  Arms: Intervention group

SUMMARY:
The main objective:

To determine the effectiveness of a treatment that combines the application of a functional upper limb orthosis together with a home-based program of specific tasks in children with unilateral cerebral palsy versus a home-based program of specific tasks in improving structure and function, activity and participation.

Hypothesis:

The application of a functional upper limb orthosis together with a home-based program of specific tasks in children with unilateral cerebral palsy results in a greater improvement in structure and function, activity and participation compared to the implementation of a home-based specific task program.

DETAILED DESCRIPTION:
Randomized clinical trial with blinding of the evaluator and the person analyzing the data.

A home-based protocol of specific tasks will be performed in both groups and one of the groups will also receive a treatment with upper limb splinting. The assessment will be made by a single evaluator with 10 years of experience in the treatment of children with motor disabilities.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of unilateral cerebral palsy (hemiplegia-hemiparesis).
2. Ages between 5 and 12 years.
3. Levels I-III of the Manual Ability Classification System (MACS)
4. Levels I-III of the Gross Motor Function Classification System (GMFCS)
5. Able to understand and respond to verbal instructions.

Exclusion Criteria:

1. Cognitive impairment identified by the school report.
2. Hand orthopedic surgery in the last 6 months.
3. Neuropharmacological intervention in the last 6 months.
4. Allergy to upper limb orthosis material.
5. Affectation of the manual function not due to the neurological condition (trauma, burn ...).
6. Current treatments not compatible with the study.
7. Other significant neurological affections (crisis, severe visual impairment ...).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Primary Outcome_Change from baseline Assisting Hand Assessment measure. Measurement of bimanual performance in pre-established tasks | Pre-intervention; Post-intervention (6 weeks after); Follow up (8 weeks after the intervention).
  Activity measurement: Assisting Hand Assessment. Measurement of bimanual performance in pre-established tasks. It quantifies the effectiveness with which the child uses his affected hand in bimanual activities.
Primary Outcome_2. Change from baseline Children's Hand-use Experience Questionnaire measure. Measurement of bimanual performance in activities of daily living. | Pre-intervention; Post-intervention (6 weeks after); Follow up (8 weeks after the intervention).
  Participation and activity measurement: Children's Hand-use Experience Questionnaire. The objective of the questionnaire is to measure bimanual performance in activities of daily living.

SECONDARY OUTCOMES:
Secondary Outcome_Change from baseline Box and Blocks Test measure. Measurement of unilateral gross manual dexterity. | Pre-intervention; Post-intervention (6 weeks after); Follow up (8 weeks after the intervention).
  Activity measurement: Box and Blocks Test assesses unilateral gross manual dexterity.
Secondary Outcome_2. Change from baseline Jebsen Hand Function Test measure. Measurement of a broad range of uni-manual hand functions required for activities of daily living. | Pre-intervention; Post-intervention (6 weeks after); Follow up (8 weeks after the intervention).
  Participation measurement: Jebsen Hand Function Test. The objective of this test is to assess a broad range of uni-manual hand functions required for activities of daily living.7 activities performed with the affected hand and healthy hand separately.
Secondary Outcome_3. Change from baseline House Thumb in Palm Deformity Classification. Classify the deformity level of thumb. | Pre-intervention; Post-intervention (6 weeks after); Follow up (8 weeks after the intervention).
  Structure and function measurement: House Thumb in Palm Deformity Classification. This tool classify the deformity levels taking into account the structure of the thumb.
Secondary Outcome_4. Change from baseline Neurological Hand Deformity Classification. This tool classify the deformity levels of wrist and fingers. | Pre-intervention; Post-intervention (6 weeks after); Follow up (8 weeks after the intervention).
  Structure and function measurement: Neurological Hand Deformity Classification. This tools classify the deformity levels taking into account the wrist, fingers.
Secondary Outcome_5. Change from baseline Grip and Pinch Strength measure. Measurement of pinch, wrist and foream strength. | Pre-intervention; Post-intervention (6 weeks after); Follow up (8 weeks after the intervention).
  Structure and function measurement: Grip and Pinch Strength. One will be used to Assess the grip of the thumb (Pinch Gauge Dynamometer) and another to assess the strength of the wrist and forearm (Hand and Wrist Dynamometer).

CONTACTS AND LOCATIONS:
Overall Officials: María Ortiz Lucas, PhD, Study Director — Universidad San Jorge; Vanesa Abuín Porras, PhD, Study Director — Universidad Europea de Madrid; Patricia Roldán Pérez, MSc, Principal Investigator — Universidad San Jorge
Locations (2):
- Spain (2):
  - AIDIMO Asociación para la investigación en la discapacidad motriz, Zaragoza
  - Universidad San Jorge, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Steenbergen B, Gordon AM. Activity limitation in hemiplegic cerebral palsy: evidence for disorders in motor planning. Dev Med Child Neurol. 2006 Sep;48(9):780-3. doi: 10.1017/S0012162206001666. PMID 16904028
- [Background] Arner M, Eliasson AC, Nicklasson S, Sommerstein K, Hagglund G. Hand function in cerebral palsy. Report of 367 children in a population-based longitudinal health care program. J Hand Surg Am. 2008 Oct;33(8):1337-47. doi: 10.1016/j.jhsa.2008.02.032. PMID 18929198
- [Background] Malagon Valdez J. [Cerebral palsy]. Medicina (B Aires). 2007;67(6 Pt 1):586-92. Spanish. PMID 18422084
- [Background] Kolb B, Whishaw IQ. Neuropsicología humana: Ed. Médica Panamericana; 2006.
- [Background] Cioni G, Sales B, Paolicelli PB, Petacchi E, Scusa MF, Canapicchi R. MRI and clinical characteristics of children with hemiplegic cerebral palsy. Neuropediatrics. 1999 Oct;30(5):249-55. doi: 10.1055/s-2007-973499. PMID 10598836
- [Background] Robaina-Castellanos GR, Riesgo-Rodriguez S, Robaina-Castellanos MS. [Definition and classification of cerebral palsy: a problem that has already been solved?]. Rev Neurol. 2007 Jul 16-31;45(2):110-7. Spanish. PMID 17642051
- [Background] Himmelmann K, Uvebrant P. The panorama of cerebral palsy in Sweden. XI. Changing patterns in the birth-year period 2003-2006. Acta Paediatr. 2014 Jun;103(6):618-24. doi: 10.1111/apa.12614. Epub 2014 Mar 24. PMID 24575788
- [Background] Pueyo-Benito R, Vendrell-Gomez P, Bargallo-Alabart N, Mercader-Sobreques JM. [Neuroimaging and cerebral palsy]. Rev Neurol. 2002 Sep 1-15;35(5):463-9. Spanish. PMID 12373681
- [Background] Burtner PA, Poole JL, Torres T, Medora AM, Abeyta R, Keene J, Qualls C. Effect of wrist hand splints on grip, pinch, manual dexterity, and muscle activation in children with spastic hemiplegia: a preliminary study. J Hand Ther. 2008 Jan-Mar;21(1):36-42; quiz 43. doi: 10.1197/j.jht.2007.08.018. PMID 18215750
- [Background] Koman LA, Gelberman RH, Toby EB, Poehling GG. Cerebral palsy. Management of the upper extremity. Clin Orthop Relat Res. 1990 Apr;(253):62-74. PMID 2180605
- [Background] Novak I, Cusick A, Lannin N. Occupational therapy home programs for cerebral palsy: double-blind, randomized, controlled trial. Pediatrics. 2009 Oct;124(4):e606-14. doi: 10.1542/peds.2009-0288. Epub 2009 Sep 21. PMID 19770175
- [Background] Elliott C, Reid S, Hamer P, Alderson J, Elliott B. Lycra((R)) arm splints improve movement fluency in children with cerebral palsy. Gait Posture. 2011 Feb;33(2):214-9. doi: 10.1016/j.gaitpost.2010.11.008. Epub 2010 Dec 4. PMID 21131201
- [Background] Ozer K, Chesher SP, Scheker LR. Neuromuscular electrical stimulation and dynamic bracing for the management of upper-extremity spasticity in children with cerebral palsy. Dev Med Child Neurol. 2006 Jul;48(7):559-63. doi: 10.1017/S0012162206001186. PMID 16780624
- [Background] Morris C. A review of the efficacy of lower-limb orthoses used for cerebral palsy. Dev Med Child Neurol. 2002 Mar;44(3):205-11. doi: 10.1017/s0012162201001943. No abstract available. PMID 12005323
- [Background] Louwers A, Beelen A, Holmefur M, Krumlinde-Sundholm L. Development of the Assisting Hand Assessment for adolescents (Ad-AHA) and validation of the AHA from 18 months to 18 years. Dev Med Child Neurol. 2016 Dec;58(12):1303-1309. doi: 10.1111/dmcn.13168. Epub 2016 Jun 13. PMID 27291981
- [Background] Holmefur M, Aarts P, Hoare B, Krumlinde-Sundholm L. Test-retest and alternate forms reliability of the assisting hand assessment. J Rehabil Med. 2009 Nov;41(11):886-91. doi: 10.2340/16501977-0448. PMID 19841839
- [Background] Holmefur M, Krumlinde-Sundholm L, Eliasson AC. Interrater and intrarater reliability of the Assisting Hand Assessment. Am J Occup Ther. 2007 Jan-Feb;61(1):79-84. doi: 10.5014/ajot.61.1.79. PMID 17302108
- [Background] Eliasson AC, Krumlinde-Sundholm L, Rosblad B, Beckung E, Arner M, Ohrvall AM, Rosenbaum P. The Manual Ability Classification System (MACS) for children with cerebral palsy: scale development and evidence of validity and reliability. Dev Med Child Neurol. 2006 Jul;48(7):549-54. doi: 10.1017/S0012162206001162. PMID 16780622
- [Background] Ohrvall AM, Krumlinde-Sundholm L, Eliasson AC. The stability of the Manual Ability Classification System over time. Dev Med Child Neurol. 2014 Feb;56(2):185-9. doi: 10.1111/dmcn.12348. Epub 2013 Nov 25. PMID 24417511
- [Background] Rosenbaum PL, Palisano RJ, Bartlett DJ, Galuppi BE, Russell DJ. Development of the Gross Motor Function Classification System for cerebral palsy. Dev Med Child Neurol. 2008 Apr;50(4):249-53. doi: 10.1111/j.1469-8749.2008.02045.x. Epub 2008 Mar 1. PMID 18318732
- [Background] Palisano RJ, Cameron D, Rosenbaum PL, Walter SD, Russell D. Stability of the gross motor function classification system. Dev Med Child Neurol. 2006 Jun;48(6):424-8. doi: 10.1017/S0012162206000934. PMID 16700931
- [Background] House JH, Gwathmey FW, Fidler MO. A dynamic approach to the thumb-in palm deformity in cerebral palsy. J Bone Joint Surg Am. 1981 Feb;63(2):216-25. PMID 7462278
- [Background] Georgiades M, Elliott C, Wilton J, Blair E, Blackmore M, Garbellini S. The Neurological Hand Deformity Classification for children with cerebral palsy. Aust Occup Ther J. 2014 Dec;61(6):394-402. doi: 10.1111/1440-1630.12150. Epub 2014 Aug 29. PMID 25169815
- [Background] Mathiowetz V, Wiemer DM, Federman SM. Grip and pinch strength: norms for 6- to 19-year-olds. Am J Occup Ther. 1986 Oct;40(10):705-11. doi: 10.5014/ajot.40.10.705. PMID 3777107
- [Background] Hepping AM, Ploegmakers JJ, Geertzen JH, Bulstra SK, Stevens M. The Influence of Hand Preference on Grip Strength in Children and Adolescents; A Cross-Sectional Study of 2284 Children and Adolescents. PLoS One. 2015 Nov 23;10(11):e0143476. doi: 10.1371/journal.pone.0143476. eCollection 2015. PMID 26599429
- [Background] Mathiowetz V, Federman S, Wiemer D. Box and block test of manual dexterity: norms for 6-19 year olds 52(5):241-5, 1985.
- [Background] Jongbloed-Pereboom M, Nijhuis-van der Sanden MW, Steenbergen B. Norm scores of the box and block test for children ages 3-10 years. Am J Occup Ther. 2013 May-Jun;67(3):312-8. doi: 10.5014/ajot.2013.006643. PMID 23597689
- [Background] Amer A, Eliasson AC, Peny-Dahlstrand M, Hermansson L. Validity and test-retest reliability of Children's Hand-use Experience Questionnaire in children with unilateral cerebral palsy. Dev Med Child Neurol. 2016 Jul;58(7):743-9. doi: 10.1111/dmcn.12991. Epub 2015 Nov 26. PMID 26610725
- [Background] Skold A, Hermansson LN, Krumlinde-Sundholm L, Eliasson AC. Development and evidence of validity for the Children's Hand-use Experience Questionnaire (CHEQ). Dev Med Child Neurol. 2011 May;53(5):436-42. doi: 10.1111/j.1469-8749.2010.03896.x. Epub 2011 Mar 17. PMID 21413973
- [Background] Jebsen RH, Taylor N, Trieschmann RB, Trotter MJ, Howard LA. An objective and standardized test of hand function. Arch Phys Med Rehabil. 1969 Jun;50(6):311-9. No abstract available. PMID 5788487
- [Background] Sears ED, Chung KC. Validity and responsiveness of the Jebsen-Taylor Hand Function Test. J Hand Surg Am. 2010 Jan;35(1):30-7. doi: 10.1016/j.jhsa.2009.09.008. Epub 2009 Dec 2. PMID 19954898
- [Derived] Roldan-Perez P, Abuin-Porras V, Buesa-Estellez A, Ortiz-Lucas M. Functional Splinting efficacy in a Specific Task Home Program for Children with Cerebral Palsy. A Randomized Controlled Trial. Dev Neurorehabil. 2022 Oct;25(7):469-478. doi: 10.1080/17518423.2022.2099027. Epub 2022 Jul 13. PMID 35822931